CLINICAL TRIAL: NCT01009645
Title: The Effect of Fact Versus Myth Messages on Receipt of Influenza Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Fact versus Myth Messages; 1R21AG031470-01 (NIH)
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Results first posted 2012-09-18 (Estimated); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Influenza Vaccination
Keywords: education; vaccination; preventive service; Prevention & Control
MeSH Terms: conditions — Influenza, Human | interventions — SUPT16H protein, human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fact Only (Experimental): The educational message used will contain facts only.
  Interventions: Behavioral: Fact Only Education Message
- Fact and Myth (Experimental): The educational material seen by this arm will contain facts and myths only.
  Interventions: Behavioral: Fact and Myth Educational Message
- Fact, Myth, Why (Experimental): The educational material seen by this arm will contain myths, facts, and refutations of the myths.
  Interventions: Behavioral: Fact, Myth, Why Educational Message
- Control (Placebo Comparator): This arm will receive fact/myth educational materials originally developed and used by the CDC.
  Interventions: Behavioral: Control Educational Message

INTERVENTIONS:
Behavioral: Fact Only Education Message — Participants randomized to this intervention will receive an educational brochure listing the facts of the influenza vaccine.
  Other Names: Fact Only
  Arms: Fact Only
Behavioral: Fact and Myth Educational Message — Participants randomized to this intervention will receive an educational brochure listing the facts and myths of the influenza vaccine.
  Other Names: Fact & Myth
  Arms: Fact and Myth
Behavioral: Fact, Myth, Why Educational Message — Participants randomized to this intervention will receive an educational brochure listing the facts, myths, and refutation of the myths of the influenza vaccine.
  Other Names: Fact, Myth, Why
  Arms: Fact, Myth, Why
Behavioral: Control Educational Message — Participants randomized to this intervention will receive an educational brochure created and used by the CDC in a previous influenza season.
  Other Names: Control
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate whether message design of educational materials increases vaccination rates among participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a scheduled appointment at least 6 weeks in advance in either the GIM or Geriatrics clinics at NMFF.
* Participant must be a patient of Northwestern Medical Faculty Foundation.
* Participant does not intend to receive the influenza vaccine.

Exclusion Criteria:

* Participant has a diagnosis of Alzheimer's Disease or Dementia
* Participant has received an influenza vaccination during either the last influenza season or the current.
* The scheduled visit is the participant's first time being seen by this doctor (appointment is to establish care in the clinic).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2009-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Medical Faculty Foundation General Internal Medicine and Geriatric Clinics, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants had scheduled appointments in a private medical clinic during October 2009 - March 2010. Potential participants were sent an opt-out letter indicating that they would be receiving a phone call to invite them to participate in a study if interested; those not opting out were contacted and asked to participate.
Pre-assignment Details: If potential participants had already received the seasonal influenza vaccination for 2009 - 2010 or responded on the phone that they "definitely intended" to receive the vaccine, they were excluded from the study. These screening questions were asked prior to enrollment into the study.
Period: Overall Study
Arm/Group | Fact Only | Fact and Myth | Fact, Myth, Why | Control
Started | 31 | 31 | 32 | 31
Completed | 29 | 23 | 28 | 26
Not Completed | 2 | 8 | 4 | 5
Not completed — Lost to Follow-up | 2 | 8 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fact Only | Fact and Myth | Fact, Myth, Why | Control | Total
Number analyzed (Participants) | 31 | 31 | 32 | 31 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 20 | 23 | 16 | 77
  >=65 years | 13 | 11 | 9 | 15 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (11.27) | 61.13 (7.46) | 63.34 (9.64) | 65.35 (8.40) | 63.16 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 23 | 24 | 98
  Male | 4 | 7 | 9 | 7 | 27
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 32 | 31 | 125

OUTCOME MEASURES:

1. Primary Outcome: Influenza Vaccination
Description: The primary outcome is receipt of influenza vaccination at appointment directly following the post-test. A pre-test was completed by participants during a telephone interview that occurred approximately two weeks prior to a scheduled clinic appointment. The post-test was completed via an in-person interview by participants immediately prior to their scheduled appointment. That is, the participants met with the Research Assistant, completed the post-test, and then proceeded to see their physician for a previously scheduled office visit.
Time Frame: 1 week following randomization
Measure: Number; unit: participants
Arm/Group | Fact Only | Fact and Myth | Fact, Myth, Why | Control
Number analyzed (Participants) | 31 | 31 | 32 | 31
participants | 4 | 1 | 3 | 4
Statistical Analysis 1: Comparison: Fact Only vs Fact and Myth vs Fact, Myth, Why vs Control; Contrast analysis was used to assess difference in vaccination status. The first contrast assessed whether or not the three newly created messages (Fact Only (FO), Fact/Myth (FM), and Fact/Myth/Refutation (FMR)) were as a group significantly different than the control message; Test type: Superiority or Other; p < 0.05, Contrast Analysis — The a priori threshold for statistical significance was p <0.0167 as the p-value was adjusted for multiple comparisons (three planned contrasts); Bonferroni correction used (3 planned contrasts)
Statistical Analysis 2: Comparison: Fact Only vs Fact and Myth vs Fact, Myth, Why; Contrast analysis was used to assess difference in vaccination status. The second contrast assessed whether the FO and FMR conditions were significantly different from the FM message; Test type: Superiority or Other; p < 0.05, Contrast Analysis — [p-value comment as in outcome 1, analysis 1]; Bonferroni correction used (3 planned contrasts)
Statistical Analysis 3: Comparison: Fact Only vs Fact, Myth, Why; Contrast analysis was used to assess difference in vaccination status. The third contrast assessed whether the FO and the FMR message conditions were significantly different; Test type: Superiority or Other; p < 0.05, Contrast Analysis — [p-value comment as in outcome 1, analysis 1]; Bonferroni correction used (3 planned contrasts)

2. Secondary Outcome: Recall Accuracy
Description: Participants were given 8 statements about the flu/flu shot and asked to recall if they had seen the statement on the message they received via FedEx. Participants responded that statement had been "presented as a fact," "presented as a myth," "presented, but I don't recall if it was a fact or a myth," or "not presented." Participants scored 1 for each correct answer; 0 for each incorrect answer or for response "I don't recall." Recall accuracy was calculated among each message format, range for recall accuracy was 0 - 8 with 0 indicating no correct answers and 8 representing 100% accuracy. Thus units of measurement are "units on a scale" to represent participant scores out of 8 on the recall items.
Time Frame: 1 week following receipt of message
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fact Only | Fact and Myth | Fact, Myth, Why | Control
Number analyzed (Participants) | 31 | 31 | 32 | 31
units on a scale | 3.13 (1.66) | 4.52 (1.96) | 5.67 (1.65) | 4.77 (1.82)
Statistical Analysis 1: Comparison: Fact Only vs Fact and Myth vs Fact, Myth, Why vs Control; Test type: Superiority or Other; p < 0.05, ANOVA; used Scheffe's post-hoc analysis

ADVERSE EVENTS:
Arm/Group | Fact Only | Fact and Myth | Fact, Myth, Why | Control
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/32 | 0/31

LIMITATIONS AND CAVEATS:
Low participation in the trial due to the emergence of H1N1; many individuals >50 years of age opted to receive seasonal flu vaccine as they were initially unable to receive the H1N1 vaccine. Hence, the available study population shrank markedly.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes